CLINICAL TRIAL: NCT05471154
Title: Non-invasive Brain Stimulation of the Prefrontal Cortex in Substance Use Disorders
Acronym: NIBSSUD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22022NIBSSUD
Record Dates: First submitted 2022-07-06; First posted 2022-07-22 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-12

CONDITIONS: Alcohol Use Disorder (AUD)
Keywords: AUD; SUD; tDCS; NIBS; craving; abstinence; EEG
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Intervention Model Description: In this study, High-Definition transcranial direct current stimulation is used as treatment/intervention (HD-tDCS). HD-tDCS will be applied with a current of 2 mA during 20 minutes. Participants are semi-randomly assigned to the two experimental groups (active stimulation vs. sham) by the coordinating researcher, taking into account the sex of the participant. The sham condition will use the same montage but stop stimulation after a short ramp-up of 1 minute).
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blind: another researcher than the one collecting data will program the codes of the ad verum vs. sham stimulation so that both participant and researcher (collecting data) are blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active HD-tDCS (Experimental): Half of all subjects will receive active HD-tDCS (randomly assigned): anodal stimulation on the right dorsolateral prefrontal cortex. Stimulation will consist of 20 minutes 2mA anodal stimulation of the right dorsolateral prefrontal cortex.
  Interventions: Device: High Definition transcranial direct current stimulation (HD-tDCS)
- Sham HD-tDCS (Sham Comparator): Half of all subjects will receive sham HD-tDCS (randomly assigned). A ramp-up of 1 minute will be used to induce the same feelings as during the active tDCS, but will then stop the stimulation. A short ramp up is repeated in the last minute of the protocol.
  Interventions: Device: High Definition transcranial direct current stimulation (HD-tDCS)

INTERVENTIONS:
Device: High Definition transcranial direct current stimulation (HD-tDCS) — HD-tDCS is used at 2mA and during 20 minutes and with electrodes positioned on regions F4 (anode), Fp2, Fz, F8 and C4 (cathodes), according to the international 10-20 electroencephalogram system. 5 sessions are given on 5 following days. The material used in this study is the Soterix Medical 1x1 tES mini-CT and HD 4x1 splitter, produced by Soterix Medical Inc., 237 W 35th St, New York, NY 10001, United States of America.

SUMMARY:
Every year, alcohol causes 3 million deaths worldwide. Even though a lot of treatments already exist, many of them are characterized by a high percentage of drop-out or relapse. Transcranial direct current stimulation (tDCS), a NIBS, is receiving increased attention as a possible new addiction treatment. However, little consensus exists in the concrete parameters (e.g. montage, current, intensity). Moreover, a lot of tDCS research focuses on subjective outcomes, like the report of craving, which are more prone to different biases and fluctuations. In this study, we aim to investigate the effect of HD-tDCS, a more focal stimulation variant, on AUDs. Using this intervention, stimulation can be restricted to one hemisphere, controlling for possible inhibition effects of the cathode. A between-subject design will be carried out, including patients with an AUD. Participants will receive 5 sessions of either real or sham right anodal HD-tDCS over the dorsolateral prefrontal cortex (dlPFC). Craving will be accounted for at baseline and after every stimulation session. Moreover, we will measure the activity of the brain in rest and during two inhibition tasks (Go/NoGo and cue reactivity task). This objective measure will be carried out both before (baseline) and at two time points after the stimulation, to measure effects on both the short and longer term. One month after the intervention, abstinence will be checked through a follow-up phone call. Through this study, we aim to describe positive effects of right dlPFC stimulation on craving, abstinence, and EEG measures.

DETAILED DESCRIPTION:
Population

This study will focus on patients with AUD, as these are the easiest to recruit. Participants in this study will be enrolled in a residential SUD treatment or a day hospital SUD treatment. As such, medical supervision can be guaranteed. In addition, sobriety is assessed objectively and routinely as part of TAU, enabling exclusion of patients under influence of alcohol. Cognitive impairment will be assessed using the MoCA and participants with a score below 10 (severe cognitive impairment) will be excluded.

Design

This study will use a between-subjects design. The experiment will be conducted double-blind to minimalize placebo effects and researcher bias. Group allocation will be conducted semi-randomly, with matching of participants' sex. The otherwise identical placebo protocol features sham stimulation (after a short ramp up, current drops again). The short ramp up is used to induce the same sensations as in the stimulation group (possible itching and tingling).

Measures

Self-report

Self-report measures will be collected prior to the intervention to discern endophenotypes predicting treatment response. The Behavioral Inhibition/Behavioral Activation System (BIS/BAS), Effortful Control Scales, Barrat Impulsiveness Scale and the Alcohol Use Disorders Identification Test (AUDIT) are collected. The Beck Depression Inventory (BDI) will be collected both before and after intervention.

Cognitive screening

The Montreal Cognitive Assessment (MoCA) will be used to exclude patients with severe cognitive impairment. Participants with a score of 10 or lower on the MoCA will be excluded from the study.

Medication regime

The medication regime of the participants will be registered, since medication may influence tDCS effects.

Resting state EEG

A resting state EEG is collected before the intervention as well as immediately after the first stimulation session and after the last stimulation session. These timepoints are used to collect data concerning the effect of tDCS on both short term and longer term.

ERPs and behavioral measures

Apart from resting state, event related potentials (ERP's) will be collected at the same time points, during different behavioral tasks: a cue reactivity task reflecting activation of the reward system and a Go-NoGo task reflecting executive functions, more concrete response inhibition.

* Cue-reactivity task: In this task, participants will be requested to indicate the occurrence of any infrequent stimulus by pressing the response button as fast as possible. Participants will be shown successions of pictures of a person drinking water (frequent), alcohol (infrequent) or soft drinks (equally infrequent). All stimuli will be presented in a random order. Three different alcohol-related pictures will be used, selected during the screening for alcohol preference.
* Go/NoGo task: In this task, participants have to press a button as fast as possible, whenever the Go stimulus (the letter M) is displayed. When another, infrequent stimulus is displayed (NoGo, the letter W), they have to refrain from pressing the button. The letters are superimposed on an alcohol-related picture or a non-alcohol related picture.

In both tasks, trials followed by incorrect responses will be eliminated from the data set. Reaction times and percentage of errors will be registered as behavioral measures.

Safety and blinding

After every session of HD-tDCS adverse effects will be assessed. Moreover, participants will systematically be asked whether they believe to have received real or placebo stimulation in the past session.

Subjective craving

A subjective craving measure will be carried out before the intervention and after every stimulation session.

Follow-up

1 month after the last stimulation session, verbally self-reported abstinence status will be registered. To do so, the Quick Drinking Screen (QDS) will be used.

Intervention

5 sessions of 2mA HD-tDCS (active or sham) will be used as intervention during 20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* DSM-V criteria for alohol use disorder
* dutch speaking
* 18-65 years old
* abstinence in the past 10 days

Exclusion Criteria:

* diagnosis or family history of epilepsy
* a history of severe brain injury
* a cardiac pacemaker or electronic implants
* migraine
* a scalp skin condition
* pregnancy
* concurrent treatment with benzodiazepines
* hairstyle incompatible with EEG-measurements
* a psychotic disorder or neurological disease
* severe cognitive impairment defined as a score lower than 10 on the Montreal Cognitive Assessment (MoCA).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-09-22 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
Abstinence | 1 month after the intervention
  1 month after the last stimulation session, verbally self-reported abstinence status will be registered. To do so the Quick Drinking Screen (QDS) will be used during a phone call by the researcher.

SECONDARY OUTCOMES:
ERP measures | Total estimated period of one week: pre-intervention (on day 1;T1), after a first stimulation session (day 1, 30 minutes after T1) and after the full intervention of 5 sessions (on day 5,4 days after T1)
  We will measure the ERP during a cue-reactivity and a Go/NoGo task, pre-intervention, immediately after the first stimulation session and immediately after the last stimulation session.
Craving measures | Total estimated period of one week: measure pre-intervention (day 1, T1) and after every stimulation session (T1 + 1 hour, T1 + 1 day, T1 + 2 days, T1 + 3 days and T1+ 4 days)
  subjective craving ratings on a Visual Analogue Scale (VAS), ranging from 0 to 10, 0 being no feeling of craving and 10 being very heavy feeling of craving
Effortful control scale (EC) | The week before first day of intervention (T1), during a block of questionnaires (estimated at 1 hour in time spending)
  The effortful control scale aims to assess temperamental capacity for effortful control us-ing 19 items. The items need to be rated from 1 (not applicable) to 7 (very applicable) or X (never been in this situation)
resting state EEG in alpha band | otal estimated period of one week: pre-intervention (on day 1;T1), after a first stimulation session (day 1, 30 minutes after T1) and after the full intervention of 5 sessions (on day 5,4 days after T1)
  Resting state EEG will be collected during 5 minutes. Afterwards, the power in the different frequency bands will be compared, focusing on prefrontal asymmetry in alpha power.
Behavioral inhibition system/behavioral approach system (BIS/BAS) Scale | The week before first day of intervention (T1), during a block of questionnaires (estimated at 1 hour in time spending)
  The BIS/BAS questionnaire consists of 24 items. The questionnaire aims to measure the two motivational systems: the behavioral inhibition system and the behavioral approach system. Each item needs to be rated between 1 (true/applicable for me) to 4 (not true/applicable for me)
Barratt Impulsivity Scale (BIS) | The week before first day of intervention (T1), during a block of questionnaires (estimated at 1 hour in time spending)
  the Barratt Impulsivity Scale (BIS-11) is a questionnaire that aims to assess impulsiveness as a personality construct. The Scale consists of 30 items, that need to be rated from "never/almost never" to "almost always"
Montreal Cognitive Assessment (MoCA) | The week before first day of intervention (T1), during a block of questionnaires (estimated at 1 hour in time spending)
  the MoCA will be used to exclude patients with severe cognitive impairment. It is a short cognitive screening tool, that takes around 10 minutes to complete. The question-naire consists of one page with questions, for a total amount of 30 points. The different tasks focus on short term memory recall, visuospatial abilities, executive functions, at-tention, concentration and working memory, language and orientation to time and place. A score of 26 or higher is considered normal. For exclusion, we will use the cut off of 10 (severe cognitive impairment) in the Dutch version of the MoCA
screening alcohol preference | The week before first day of intervention (T1), during a block of questionnaires (estimated at 1 hour in time spending)
  During the first meeting, participants will be shown pictures of various alcoholic drinks. Participants will be asked to rank these pictures based on how strong the craving they elicit. The highest ranked stimuli will be used in the behavioral / ERP tasks.
Alcohol Use Disorders Identification Test (AUDIT) | The week before first day of intervention (T1), during a block of questionnaires (estimated at 1 hour in time spending)
  the AUDIT will be used to measure and objectify the severity of the participants' alcohol problem. The questionnaire consists of 10 questions and covers the domains of drinking behavior, alcohol consumption and alcohol-related problems. Questions need to be answered by indicating a value between 0 (Never/No/Few) and 4 (Daily/Yes/Almost daily)
Beck Depression Inventory (BDI) | The week before first day of intervention (T1) and after intervention (T2)
  the BDI will be used to measure depression and depressive symptoms. The questionnaire consists of 21 items aiming to measure symptoms like irritability, physical symptoms and helplessness.

CONTACTS AND LOCATIONS:
Overall Officials: Natacha Deroost, PhD, Study Chair — Vrije Universiteit Brussel; Kris Baetens, PhD, Study Director — Vrije Universiteit Brussel; Geert Dom, MD, Study Chair — PC Multiversum Boechout; Marianne Destoop, MD, Study Chair — PC Multiversum Boechout
Locations (1):
- Multiversum, Boechout, Antwerpen, Belgium

IPD SHARING:
Plan to Share IPD: No